CLINICAL TRIAL: NCT03676647
Title: Retrospective-Prospective Collection of Thyroid Specimens After FNA
Brief Title: Diagnostic DNA Methylation Signature in Diagnosing Thyroid Cancer After Fine-Needle Aspiration in Patients With Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18077; NCI-2018-01910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18077 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Gland Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — DDMS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Diagnostic DNA Methylation Signature in Diagnosing Thyroid Cancer After Fine-Needle Aspiration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (biospecimen collection): Previously collected FNA aspiration specimen samples are analyzed via DDMS assay. Participants undergo FNA aspiration for collection of tissue samples for analysis via DDMS assay.
  Interventions: Other: Diagnostic DNA Methylation Signature

INTERVENTIONS:
Other: Diagnostic DNA Methylation Signature — Undergo collection of tissue samples
  Other Names: DDMS

SUMMARY:
This trial studies how well the diagnostic deoxyribonucleic acid (DNA) methylation signature works in detecting thyroid cancer in patients with thyroid nodules. Using diagnostic testing, such as the diagnostic DNA methylation signature, may be a less invasive way to check for thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate a novel epigenetic thyroid nodule diagnostic test, diagnostic DNA methylation signature (DDMS) in a retrospective-prospective study with leftover of fine needle aspiration biopsies.

OUTLINE:

Previously collected FNA aspiration specimen samples are analyzed via DDMS assay. Participants undergo FNA aspiration for collection of tissue samples for analysis via DDMS assay.

After completion of study, patients are followed up yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing FNA for thyroid nodule diagnosis.
* Any race and ethnicity are eligible for the study.
* Patient should have thyroid nodule(s) with indeterminate diagnosis after FNA (Bethesda category of indeterminate FNA [III-V]).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People undergoing fine needle aspiration.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the diagnostic deoxyribonucleic acid (DNA) methylation signature (DDMS) | Up to 5 years
  Will be assessed by taking the ratio of the number of thyroid cancer specimens diagnosed as cancer using the DDMS and the total number of thyroid cancer specimens according to the final diagnosis. Will determine the 95% confidence intervals.
Specificity of DDMS | Up to 5 years
  Will be assessed by taking the ratio of the number of benign nodules diagnosed by DDMS and the total number of benign thyroid nodule specimens according to the final diagnosis. Will determine the 95% confidence intervals.
Positive predictive value (PPV) | Up to 5 years
  Will calculate PPV by dividing the number of true thyroid cancer specimens by the number of thyroid cancer diagnosis by DDMS. Will determine the 95% confidence intervals.
Negative predictive value (NPV) | Up to 5 years
  Will calculate NPV by dividing the number of benign nodules by the number of benign diagnosis by DDMS. Will determine the 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hahn, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States